CLINICAL TRIAL: NCT05855330
Title: Prospective Open-Label Pilot Study of Arginine Replacement Therapy in Children Hospitalized With COVID-19
Brief Title: Arginine Replacement Therapy in COVID-19
Acronym: ART-COVID19
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Claudia R. Morris, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005572
Record Dates: First submitted 2023-05-09; First posted 2023-05-11 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- L-arginine loading dose + standard dose (Active Comparator): L-arginine loading dose (200 mg/kg IV) + standard dose (100 mg/kg IV TID).
  Interventions: Drug: Arginine Hydrochloride
- Standard dose (Active Comparator): Standard dose (100mg/kg IV TID).
  Interventions: Drug: Arginine Hydrochloride
- Low dose (Active Comparator): Low dose (25mg/kg IV TID).
  Interventions: Drug: Arginine Hydrochloride

INTERVENTIONS:
Drug: Arginine Hydrochloride — Arginine will be infused based on the manufacturer's instructions (R-Gene 10, Pfizer), over 30 minutes. However, rates may be slowed to over 60 minutes for patients experiencing symptoms of flushing, nausea, vomiting, or headache at the research team's discretion. Pediatric doses will be drawn up by the pharmacy.
  Other Names: L-arginine

SUMMARY:
This study aims to investigate if receiving doses of arginine (a protein in the body) will improve mitochondria function in children with COVID-19.

The study will be performed at the Children's Healthcare of Atlanta, Arthur M. Blank Hospital. Patients will be randomized to receive one of three doses of arginine three times a day for five days or at discharge whichever comes first.

DETAILED DESCRIPTION:
In the early stages of COVID-19, it was believed that children were immune or had very mild disease. Given the unfolding pandemic, children's cases are exhibiting an increasing global trend and are associated with some serious complications in addition to more long-term complications such as multisystem inflammatory syndrome in children (MIS-C) and "Long Covid". A significant number of hospitalized and critically ill pediatric patients have now been documented, in addition to a high number of emergency department (ED) visits despite previous reports suggesting rare or mild disease in children. The research team and others have shown that severe COVID-19 and MIS-C are associated with acute arginine deficiency in both adults and children. There has been increased evidence of the role of the endothelium associated with severe inflammation in COVID-19. Low plasma arginine bioavailability has been implicated in endothelial dysfunction, immune regulation, and hypercoagulation. The research team also identified high sPLA2 levels in COVID-19 and MIS-C, an observation previously made in children with Kawasaki's Disease. Subsequent studies have shown that sPLA2 is associated with the pathobiology leading to COVID-19 mortality, with enzyme levels 10-fold higher in people who died vs. mild disease, and is also associated with Mito dysfunction. Not only could sPLA2 represent a prognostic indicator of disease severity, but it also represents a mechanism with potential therapeutic targets.

Information learned from the Mito activity in COVID-19 can contribute to further understanding of severe acute respiratory syndrome by coronavirus (SARS-CoV-2) infection. This data may help guide future treatment targets and strategies.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of COVID-19 requiring admission to the hospital for treatment of COVID-19 infection
* Age 3 years - 21 years of age

Exclusion Criteria:

* Severe hepatic dysfunction: ALT> 6 x Upper limit of normal
* Renal dysfunction: Creatinine > 1.5 x upper limit of normal or on dialysis
* Acute Stroke
* Pregnancy
* Allergy to arginine
* Past history of severe cardiac disease or significant cardiac surgery [minor procedures like ventricular septal defect (VSD) repair are not an exclusion]
* History of significant pulmonary disease [Cystic Fibrosis, sickle cell disease (SCD)]
* History of organ transplant
* History of metabolic or mitochondrial disease (including Diabetes)
* History of severe neurocognitive delays (severe cerebral palsy, anoxic brain injury)
* History of ventriculoperitoneal (VP) shunt or hydrocephalus
* PI discretion that the patient is not an ideal candidate for the study
* History of HIV of immune compromise

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in mitochondrial function | Baseline and day 5
  Complex-IV activity changes will be measured to estimate mitochondrial function before and after administration for L-arginine

SECONDARY OUTCOMES:
Change in amino acids | Baseline and day 5
  arginine (ARG) ornithine (ORN) and citrulline (CIT) will be measured before and after administration for L-arginine
Change in the arginase-1 activity/concentration | Baseline and day 5
  arginase-1 will be measured before and after administration for L-arginine
Change in myeloid-derived suppressor cells (MDSC-source of arginase-1) | Baseline and day 5
  Myeloid-derived suppressor cells (MDSC) producing arginase-1 will be measured in the peripheral blood before and after administration of L-arginine
Change in the level of cytokines (IL-6) | Baseline and day 5
  Cytokines are biomarkers for inflammation. Cell supernatants will be collected and analyzed for different cytokines.
Change on secretory phospholipase (sPLA2). | Baseline and day 5
  Serum activity of secretory phospholipase (sPLA2) will be measured before and after administration for L-arginine

CONTACTS AND LOCATIONS:
Overall Officials: Claudia R. Morris, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta (CHOA), Arthur M. Blank, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request, the research team will share de-identified data with researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data are available for at least 5 years after publication of primary results.
Access Criteria: Data are available for at least 5 years, available upon request from PI, directed to claudia.r.morris@emory.edu